CLINICAL TRIAL: NCT02862158
Title: Evaluation of Different Frequency Doubling Technology (FDT) Mobile Devices for Visual Field Assessment
Brief Title: Frequency Doubling Technology (FDT) Mobile Visual Field Testing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Richard K. Lee, Associate Professor of Ophthalmology, Cell Biology and Neuroscience Graduate Program, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20150968
Record Dates: First submitted 2016-07-18; First posted 2016-08-10 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): FDT visual field will be compared to standard HVF in detecting glaucomatous visual field loss
  Interventions: Device: FDT visual field; Device: Standard HVF

INTERVENTIONS:
Device: FDT visual field
Device: Standard HVF

SUMMARY:
This is a single center, prospective study to evaluate the efficacy and reproducibility of frequency doubling technology (FDT)-based visual field devices compared to conventional Humphrey Visual Field (HVF) perimetry. The investigators plan to enroll 500 patients in this study.

DETAILED DESCRIPTION:
Glaucoma is a leading cause of irreversible and preventable blindness world-wide. Insufficient evidence exists to support routine screening for glaucoma in a primary care setting due to the relatively low prevalence of the disease (Guirguis-Blake, 2005 and Moyer, 2013). Frequency doubling technology (FDT)-based perimetry is a relatively inexpensive and portable visual field testing device with a short testing time that has shown reasonable efficacy, sensitivity and specificity in screening for glaucoma in clinic- and community-based settings (Mansberger, 2005 and Nomoto 2009).

The aim of our study is to compare the efficacy and reproducibility of FDT perimetry platforms compared with Humphrey Visual Field (HVF) perimetry (which is the gold clinical standard in clinics and hospitals) in detecting glaucomatous visual field defects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 and over) who speak English, Spanish or Creole, and are capable of providing informed consent and who have a Humphrey Visual Field (HVF) test within the prior the 6 months preceding enrollment are eligible for enrollment in this non-invasive study. Patients will be recruited from among patients at the Bascom Palmer Eye Institute clinics during their regularly scheduled clinic visits. No advertising will be used to recruit patients.

Exclusion Criteria:

* Adults unable to consent, individuals who are not yet adults (infants, children and teenagers), pregnant women and prisoners and other vulnerable populations will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-08; Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Pattern of visual field loss in FDT visual fields as compared with standard HVF | The investigators anticipate to enroll the subjects over a period of 12 months. The estimated time required for data analysis is 6 months following enrollment of all subjects.
  Visual Field

SECONDARY OUTCOMES:
Mean deviation (MD) in FDT visual fields as compared with standard HVF | The investigators anticipate to enroll the subjects over a period of 12 months. The estimated time required for data analysis is 6 months following enrollment of all subjects.
  Visual Field
Pattern standard deviation (PSD) in FDT visual fields as compared with standard HVF | The investigators anticipate to enroll the subjects over a period of 12 months. The estimated time required for data analysis is 6 months following enrollment of all subjects.
  Visual Field

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lee, MD, PhD, Principal Investigator — University of Miami / Bascom Palmer Eye Institute
Locations (1):
- Bascom Palmer Eye Institute, University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guirguis-Blake J. Rationale for the USPSTF recommendation on screening for glaucoma. Am Fam Physician. 2005 Oct 1;72(7):1184, 1187. No abstract available. PMID 16225022
- [Background] Moyer VA; U.S. Preventive Services Task Force. Screening for glaucoma: U.S. Preventive Services Task Force Recommendation Statement. Ann Intern Med. 2013 Oct 1;159(7):484-9. doi: 10.7326/0003-4819-159-6-201309170-00686. PMID 24325017
- [Background] Mansberger SL, Johnson CA, Cioffi GA, Choi D, Krishnadas SR, Srinivasan M, Balamurugan V, Kim U, Smith SD, Wilkins JH, Gritz DC. Predictive value of frequency doubling technology perimetry for detecting glaucoma in a developing country. J Glaucoma. 2005 Apr;14(2):128-34. doi: 10.1097/01.ijg.0000151883.07232.54. PMID 15741814
- [Background] Nomoto H, Matsumoto C, Takada S, Hashimoto S, Arimura E, Okuyama S, Shimomura Y. Detectability of glaucomatous changes using SAP, FDT, flicker perimetry, and OCT. J Glaucoma. 2009 Feb;18(2):165-71. doi: 10.1097/IJG.0b013e318179f7ca. PMID 19225357